CLINICAL TRIAL: NCT02277340
Title: Endoscopic Treatment of Pilonidal Sinus May Decrease the Recurrence After Crystallized Phenol Application
Brief Title: Endoscopic Pilonidal Sinus Treatment With Additional Crystalized Phenol
Acronym: EPSITCRYSP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, I Ethem Gecim, Prof Dr, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRKAP-001
Record Dates: First submitted 2014-10-02; First posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EAPA for Pilonidal Disease (Experimental): The abbrevition EAPA is used to describe the study. The cohort of pilonidal disease patients treated who do not have an acute abscess or other problems like hydradenitis suppurativa, has been treated by endoscopy assisted fulguration of the inner surface and additional crystallized phenol application for further clean up of the remaining tissue as well as preventing bacterial growth.
  Interventions: Procedure: EAPA

INTERVENTIONS:
Procedure: EAPA — Under sedation and local anesthesia, a pit of pilonidal disease is widened, hair and debris removed and cavity first ablated by endoscopy assisted diathermy the filled with crystallized phenol. The remaining pits were also fulgurated.

SUMMARY:
This study presents 23 sacrococcygeal pilonidal disease cases treated with endoscopic cleaning and fulguration of pilonidal sinus inner surfaca followed by application of crystallized phenol into the sinus.

DETAILED DESCRIPTION:
Endoscopic treatment and crytallized phenol application are two sovereign treatments described for pilonidal disease. The curative rate may be as low as 65 % and the recurrence rate is at least 10 % after crystallized phenol alone application for pilonidal disease. The experience with endoscopic treatment of pilonidal sinus is only limited but at least 4 % recurrence rate was reported.

In this study a preliminary group of 23 patients were treated with combination of these two modalities between February to May 2014 and at the end of 6-9 months follow up, there was no recurrence after excellent cosmetic results. Patients were all operated and mild sedation and local anesthesia. There was no serious complication but only some skin irritation was noticed secondary to phenol burn. Some patients felt mild pain and the pain was self limited in most cases where only a few needed oral pain killers. Some patients were observed to have mild drainage from the sinus but only two of them needed further application of phenol crystals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pilonidal disease with no acute abscess

Exclusion Criteria:

* Patients with aacute pilonidal disease abscess

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Endoscopic Pilonidal Sinus Treatment With Additional Crystalized Phenol Application | six months
  "Number of Participants with Adverse Events as a Measure of Safety and Tolerability".

SECONDARY OUTCOMES:
Endoscopic Pilonidal Sinus Treatment With Additional Crystalized Phenol Application | six months
  Number of Participants without healing of the sinus.
Endoscopic Pilonidal Sinus Treatment With Additional Crystalized Phenol Application | six months
  Recurrence rate

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim E Gecim, MD, Study Chair — Professor of Surgery, Ankara University Medical School